CLINICAL TRIAL: NCT05824585
Title: A Phase 1, Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Efficacy of DZD8586 in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (B-NHL)
Brief Title: DZD8586 in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dizal Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DZ2022B0002
Record Dates: First submitted 2023-03-30; First posted 2023-04-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DZD8586 (Experimental)
  Interventions: Drug: DZD8586

INTERVENTIONS:
Drug: DZD8586 — DZD8586 treatment starting from 50 mg once daily. If tolerated, subsequent cohorts will test increasing doses of DZD8586.

SUMMARY:
This study will treat patients with B-NHL who have relapsed, progressed, or were intolerant to systemic therapy progressed following prior therapy. This study will help to understand what type of side effects may occur with the drug treatment. It will also measure the levels of drug in the body and assess its anti-cancer activity as monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants who have provided ICF with age ≥ 18 yrs
2. ECOG performance 0-2, no deterioration in the past 2 weeks
3. Participants with relapsed or refractory B-NHL must have cytologically or histologically confirmed B-cell lymphoma
4. Adequate bone marrow reserve and organ system functions
5. Participants willing to comply with contraceptive restrictions

Exclusion Criteria:

1. Any unresolved > Grade 1 adverse event at the time of starting study treatment with the exception of alopecia.
2. Prior history of allogeneic hematopoietic stem cell transplantation
3. Stem cell transplantation, cell therapy, or gene therapy within 90 days. Approved small molecule therapy within 5 half-lives, investigational small molecule therapy within 14 days. Monoclonal antibodies and antibody-drug conjugates within 28 days Radiation therapy within 1 weeks
4. Live attenuated vaccines or viral vector vaccines within 4 weeks. Major surgery or significant traumatic injury within 4 weeks. History of stroke or intracranial hemorrhage within 6 months
5. Participants with non-CNSL presence of CNS or intraocular lymphoma lesions.
6. CNSL participants with systemic presence of lymphoma, unable to complete lumbar puncture, under systemic corticosteroids at a dose > 8 mg/day (dexamethasone equivalent dose) within 14 days or requiring immunosuppressive or biologic therapy."
7. Participants with infectious disease:
8. Clinically significant cardiac disorders or abnormalities
9. Another malignancy within 5 years prior to enrollment with the exception of adequately treated in-situ carcinoma of the cervix, uterus, basal or squamous cell carcinoma or non-melanomatous skin cancer.
10. Refractory nausea and vomiting if not controlled by supportive therapy, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption
11. Women who are breast feeding
12. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of adverse events | 30 days after the last dose, assessed up to 2 years
Part B: Objective Response Rate assessed by investigators | assessed up to 2 years

SECONDARY OUTCOMES:
Part A: Objective Response Rate assessed by investigators | assessed up to 2 years
Part A: Plasma and CSF concentration of DZD8586 | through discontinuation of treatment up to 10 weeks
Part B: Duration of Response assessed by investigators | from date of first documented response until the date of documented progression, assessed up to 2 years
Part B: Incidence of adverse events | 30 days after the last dose, assessed up to 2 years
Part B: Plasma and CSF concentration of DZD8586 | through discontinuation of treatment, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Tianwei Zhang, Study Director — Dizal Pharma
Locations (5):
- Research site, New York, New York, United States
- Australia (4):
  - Research site, Albury, New South Wales
  - Research site, Ballarat, Victoria
  - Research site, Melbourne, Victoria
  - Research site, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No